CLINICAL TRIAL: NCT04094038
Title: The Effect of Intradialytic Parenteral Nutrition on Nutritional Status and Quality of Life in Hemodialysis Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Ewout Hoorn, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDPN1; 2018-003899-13 (EudraCT Number); NL65803.078.18 (Other: Central Commission for Human Research (CCMO)); MEC-2018-1452 (Other: Erasmus MC)
Record Dates: First submitted 2019-09-12; First posted 2019-09-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: End Stage Renal Disease; Malnutrition; Sarcopenia; Hemodialysis Complication
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition; Sarcopenia | interventions — 1-((2-hydroxyethyl)amino)-2-amino-1,2-dideoxyglucose triphenyltin(IV)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intradialytic parenteral nutrition three times weekly during 16 weeks
  Interventions: Drug: Olimel N12
- Placebo (Placebo Comparator): 5% glucose three times weekly during 16 weeks
  Interventions: Drug: Glucose IV

INTERVENTIONS:
Drug: Olimel N12 — A mixture of glucose, lipids, amino acids.
  Arms: Intervention
Drug: Glucose IV — Glucose 5%
  Arms: Placebo

SUMMARY:
Protein-energy wasting (PEW), a hypercatabolic state characterized by loss of muscle mass and fuel reserves, is highly prevalent in hemodialysis patients. Nutritional status and body composition are closely linked to morbidity, mortality and quality of life. Lean tissue mass (LTM) appears to be the best read-out for the association between nutritional status and outcomes. Intradialytic parenteral nutrition (IDPN) is occasionally used with the aim to reduce loss of LTM, but its efficacy has not been established. The goal of this study is to study the effect of IDPN on changes in LTM in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing chronic hemodialysis

Exclusion Criteria:

* Life expectancy < 6 months
* Planned kidney transplant within 4 months
* Severe overhydration leading to respiratory insufficiency
* Parenteral nutrition within four weeks prior to screening
* Severe hepatic insufficiency
* Pregnancy
* Unipolar pacemaker with a very low sensitivity threshold
* Active treatment for infection
* Acute myocardial infarction
* Circulatory shock
* Hypersensitivity for any Olimel N12 ingredient or excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in lean tissue mass | 16 weeks
  Measured by body composition monitor (BCM)

SECONDARY OUTCOMES:
Skeletal muscle quality index (SMQI) | 16 weeks
  Assessed by muscle ultrasound
Change in adipose tissue mass from baseline | 16 weeks
Change in hand grip strength from baseline | 16 weeks
  Measured by hand dynamometer, expressed as percentile of reference (by age and gender)
Change in kidney disease quality of life (KDQoL-36) energy/fatigue scale from baseline | 16 weeks
  Assessed by Kidney Disease Quality of Life-36 (KDQoL-36) survey (energy/fatigue scale, 0-100, higher is better)
Change in kidney disease quality of life (KDQoL-36, overall health rating) from baseline | 16 weeks
  Assessed by Kidney Disease Quality of Life-36 (KDQoL-36) survey (0-100, higher is better)
Positive and negative affect | 16 weeks
  Assessed by Positive and Negative Affect Schedule (PANAS, 0-100, higher is better)
Change in phase angle from baseline | 16 weeks
  Assessed by Body Composition Monitor (BCM)
Change in body weight from baseline | 16 weeks
Change in serum prealbumin concentration from baseline | 16 weeks

OTHER OUTCOMES:
Subjective global assessment (SGA) | 16 weeks
  7-point scale, 7 indicates normal nutritional status, 1 indicates severe protein energy wasting
Change in serum albumin concentration | 16 weeks
Appetite | 16 weeks
  Numeric rating scale (0-10, 10 being best appetite)

CONTACTS AND LOCATIONS:
Overall Officials: Ewout J Hoorn, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided